CLINICAL TRIAL: NCT04873700
Title: Real-world Data of Moderate to Severe Inflammatory Bowel Disease (UC and CD) in Mexico: a Multicenter, Non-interventional Study to Evaluate Disease Control, Treatment Patterns, Burden of Disease and Patient Reported Outcomes
Brief Title: A Study of Moderate to Severe Inflammatory Bowel Disease, Including Ulcerative Colitis (UC) and Crohn's Disease (CD)
Acronym: RISE-MX
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IBD-5010; U1111-1262-1609 (Registry Identifier: WHO)
Record Dates: First submitted 2021-04-23; First posted 2021-05-05 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-08

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Moderate to Severe Crohn's Disease: Participants diagnosed with moderate to severe Crohn's Disease (CD) were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the IBD treatments and use of other healthcare resources related with the management of CD.
- Mild to None Crohn's Disease: Participants diagnosed with mild to none activity of CD were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the IBD treatments and use of other healthcare resources related with the management of CD.
- Moderate to Severe Ulcerative Colitis: Participants diagnosed with moderate to severe Ulcerative Colitis (UC) were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the IBD treatments and use of other healthcare resources related with the management of UC.
- Mild to None Ulcerative Colitis: Participants diagnosed with mild to none activity of UC were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the IBD treatments and use of other healthcare resources related with the management of UC.

SUMMARY:
The main aim of this study is to check the disease activity in people with moderate to severe ulcerative colitis and Crohn's disease.

Participants will complete questionnaires about their disease and quality of life on Day 1 clinic visit. They will do this during a standard scheduled appointment with their doctor. Some of this study will also involve collecting information about participants from their medical records.

DETAILED DESCRIPTION:
This is a retrospective, cross-sectional, and non-interventional study of participants with moderate to severe IBD (UC or CD). The study will have a cross-sectional evaluation on Day 1 to provide the real-world data of disease activity, treatment patterns, burden of disease and quality of life in participants with moderate to severe UC or CD.

The study will involve an additional retrospective review of medical charts of participants of previous 3 years to describe the IBD treatments and use of other healthcare resources related with the management of UC or DC.

The study will enroll approximately 335 participants. All participants will be enrolled in one observational cohort.

This multi-center trial will be conducted in Mexico. The overall time for data collection in the study will be approximately 3 years before the start of the study (Day 1).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with moderate to severe CD or UC established for at least 6 months prior to Day 1 appointment, based on clinical, endoscopic or image criteria.
2. Participants aged 18 years or older (at the time of diagnosis of moderate to severe UC or CD).

Exclusion Criteria:

1. Has indeterminate or not classified colitis.
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with moderate to severe UC or CD will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- Mexico (12):
  - Unidad de Enfermedades Reumaticas y Cronico degenerativas, Torreón, Coahuila
  - Centro De Investigacion Clinica De Alta Especialidad "Cicae", Torreón, Coahuila
  - Endoamer S.C., Guadalajara, Jalisco
  - CIMESAP Sociedad de Responsabilidad Limitada de Capital Variable, Zapopan, Jalisco
  - Hospital Medica Sur Tlalpan, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas Y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Fundacion Santos y de la Garza Evia, Monterrey, Nuevo León
  - Oncare Oncology, San Pedro Garza García, Nuevo León
  - Hospital Zambrano Hellion TecSalud, San Pedro Garza García, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
  - Torre Medica Sanatorio Toluca, Toluca
  - Arke SMO S.A. De C.V, Veracruz

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/609c23fd1f1122001e30a79f

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at approximately 12 investigative sites in Mexico from 30 August 2021 to 17 May 2022.
Pre-assignment Details: Participants with mild to none and moderate to severe inflammatory bowel disease (Ulcerative Colitis or Crohn's Disease) were enrolled in this retrospective observational study. 335 participants were enrolled, but 9 participants had insufficient data to define level of disease activity and they were not included in the analysis. All analysis and comparisons were performed considering 326 participants.
Groups:
- Moderate to Severe Crohn's Disease: Participants diagnosed with moderate to severe CD were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the inflammatory bowel disease (IBD) treatments and use of other healthcare resources related with the management of CD.
- Moderate to Severe Ulcerative Colitis: Participants diagnosed with moderate to severe UC were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the IBD treatments and use of other healthcare resources related with the management of UC.
Period: Overall Study
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Started | 43 | 52 | 42 | 189
Completed | 43 | 52 | 42 | 189
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis | Total
Number analyzed (Participants) | 43 | 52 | 42 | 189 | 326
Age, Continuous [Mean (Full Range); unit: years] | 49.5 [20 to 82] | 42.8 [21 to 81] | 43.0 [20 to 79] | 43.4 [18 to 80] | 44.67 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 33 | 19 | 114 | 191
  Male | 18 | 19 | 23 | 75 | 135
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 43 | 52 | 42 | 189 | 326

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Active CD at Day 1
Description: Percentage of participants with active CD observed, where active CD was defined as Harvey Bradshaw index (HBI) greater than or equal to (>=) 8 or Crohn's disease active index (CDAI) >=220. CDAI assessed CD based on clinical signs and symptoms such as number of liquid stools, intensity of abdominal pain, general wellbeing, presence of comorbid conditions, use of antidiarrheal, physical examination and laboratory findings. Total score ranges from 0 to 600 points. Higher score indicates more severe disease. HBI score was used to measure disease activity of CD and consisted of 5 clinical parameters: general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications. Total score is sum of individual parameters. Score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on number of liquid stools, where higher scores indicate more severe disease. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria. Data is reported for participants with active CD.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Crohn's Disease: Participants diagnosed with moderate to severe Crohn's Disease (CD) were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the inflammatory bowel disease (IBD) treatments and use of other healthcare resources related with the management of CD.
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 95
percentage of participants | 45.3 [35.3 to 55.3]

2. Primary Outcome: Percentage of Participants With Active UC at Day 1
Description: Percentage of participants with active disease UC disease will be observed, where UC is defined as 9-point Partial Mayo Score (pMayo score) >=5. The Mayo score is composed of four categories (bleeding, stool frequency, physician assessment, and endoscopic appearance) rated from 0-3 that are summed into a total score ranging from 0-12. pMayo score consists of 3 sub scores: stool frequency, rectal bleeding, and physician global assessment of disease severity, each graded from 0 to 3. These scores are summed to give a total score range of 0 to 9; where higher scores indicating more severe disease. The pMayo score when compared with the full Mayo score and categorizes UC patients as being in remission (score of 0 to 2), having mild activity (pMayo of 3 or 4) or moderate to severe activity (pMayo of >=5).
Time Frame: Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria. Data is reported for participants with active UC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ulcerative Colitis: Participants diagnosed with UC were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the IBD treatments and use of other healthcare resources related with the management of UC.
Arm/Group | Ulcerative Colitis
Number analyzed (Participants) | 231
percentage of participants | 18.2 [13.2 to 23.2]

3. Secondary Outcome: Number of Participants With CD Based on Clinical Presentation
Description: Number of participants will be reported based on the clinical presentations (location, behavior, perianal disease, achievement of ileal disease and extraintestinal manifestations for CD participants). Clinical presentations that have data for at least one participant in the below categories are reported. Data is reported for participants with CD only.
Time Frame: Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria. Data is reported for participants with CD only. Overall number analyzed is the number of participants available for analysis. Number analyzed is the number of participants with data available for each category of the clinical presentation.
Measure: Count of Participants; unit: Participants
Groups:
- Moderate to Severe Crohn's Disease: Participants diagnosed with moderate to severe Crohn's Disease (CD) were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the inflammatory bowel disease (IBD) treatments and use of other healthcare resources related with the management of CD.
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease
Number analyzed (Participants) | 7 | 30
Participants
  Location: Ileal(L1): number analyzed (Participants) | 6 | 26
  Location: Ileal(L1) | 0 | 9
  Location: L1+Isolated Upper GI Tract Disease(L4): number analyzed (Participants) | 6 | 26
  Location: L1+Isolated Upper GI Tract Disease(L4) | 0 | 1
  Location: Colonic Disease (L2): number analyzed (Participants) | 6 | 26
  Location: Colonic Disease (L2) | 1 | 5
  Location: L2 + L4: number analyzed (Participants) | 6 | 26
  Location: L2 + L4 | 1 | 0
  Location: Ileocolic(L3): number analyzed (Participants) | 6 | 26
  Location: Ileocolic(L3) | 4 | 11
  Behavior: Non stenosing/non penetrating: number analyzed (Participants) | 6 | 26
  Behavior: Non stenosing/non penetrating | 0 | 10
  Behavior: Stenosing (B2): number analyzed (Participants) | 6 | 26
  Behavior: Stenosing (B2) | 5 | 12
  Behavior: B2+Perianal Disease (P): number analyzed (Participants) | 6 | 26
  Behavior: B2+Perianal Disease (P) | 0 | 2
  Behavior: Penetrating (B3): number analyzed (Participants) | 6 | 26
  Behavior: Penetrating (B3) | 1 | 1
  Behavior: B3+P: number analyzed (Participants) | 6 | 26
  Behavior: B3+P | 0 | 1
  Perianal Disease: None: number analyzed (Participants) | 6 | 26
  Perianal Disease: None | 4 | 23
  Perianal Disease: Indolent Fistula: number analyzed (Participants) | 6 | 26
  Perianal Disease: Indolent Fistula | 0 | 3
  Perianal Disease: Active Fistula: number analyzed (Participants) | 6 | 26
  Perianal Disease: Active Fistula | 1 | 0
  Perianal Disease: Hemorrhoids: number analyzed (Participants) | 6 | 26
  Perianal Disease: Hemorrhoids | 1 | 0
  Ileal Disease: Achievement ≥1: number analyzed (Participants) | 6 | 22
  Ileal Disease: Achievement ≥1 | 3 | 19
  Ileal Disease: Achievement <1: number analyzed (Participants) | 6 | 22
  Ileal Disease: Achievement <1 | 3 | 3
  Extraintestinal Manifestations: Peripheral arthritis | 3 | 4
  Extraintestinal Manifestations: Aphthous ulcers | 0 | 2
  Extraintestinal Manifestations: Episcleritis | 0 | 1
  Extraintestinal Manifestations: Uveitis | 1 | 1
  Extraintestinal Manifestations: Osteoporosis | 0 | 1
  Extraintestinal Manifestations: Anemia | 2 | 0
  Extraintestinal Manifestations: Hematological alteration | 0 | 1
  Extraintestinal Manifestations: Other | 1 | 20
Statistical Analysis 1: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Location of disease; Test type: Superiority; p = 0.0701, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 2: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Disease behavior; Test type: Superiority; p = 0.1383, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 3: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Perianal disease; Test type: Superiority; p = 0.0478, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 4: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Ileal disease; Test type: Superiority; p = 0.1454, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 5: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Extraintestinal manifestations: Peripheral arthritis; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 6: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Extraintestinal manifestations: Aphthous ulcers; Test type: Superiority; p = 0.4992, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 7: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Extraintestinal manifestations: Episcleritis; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 8: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Extraintestinal manifestations: Uveitis; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 9: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Extraintestinal manifestations: Osteoporosis; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 10: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Extraintestinal manifestations: Anemia; Test type: Superiority; p = 0.2022, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 11: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Extraintestinal manifestations: Hematological alteration; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 12: Comparison: Moderate to Severe Crohn's Disease vs Mild to None Crohn's Disease; Extraintestinal manifestations: Other; Test type: Superiority; p = 0.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test

4. Secondary Outcome: Number of Participants With UC Based on Clinical Presentation
Description: Number of participants will be reported based on the clinical presentations (location, behavior, and extraintestinal manifestations,). Clinical presentations that have data for at least one participant in the below categories are reported. Data is reported for participants with UC only.
Time Frame: Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria. Data is reported for participants with UC only. Overall number analyzed is the number of participants available for analysis. Number analyzed is the number of participants with data available for each category of the clinical presentation.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 14 | 103
Participants
  Location - Distal UC: Proctitis(E1): number analyzed (Participants) | 14 | 98
  Location - Distal UC: Proctitis(E1) | 2 | 10
  Location - Distal UC: Proctosigmoiditis(E1): number analyzed (Participants) | 14 | 98
  Location - Distal UC: Proctosigmoiditis(E1) | 3 | 14
  Location - Left sided: Mucosa inflammation extending up to splenic flexure(E2): number analyzed (Participants) | 14 | 98
  Location - Left sided: Mucosa inflammation extending up to splenic flexure(E2) | 5 | 22
  Location - Pancolitis: Mucosa inflammation up to proximal transverse colon and beyond(E3): number analyzed (Participants) | 14 | 98
  Location - Pancolitis: Mucosa inflammation up to proximal transverse colon and beyond(E3) | 4 | 52
  Behavior - clinical remission (asymptomatic)(S0): number analyzed (Participants) | 14 | 98
  Behavior - clinical remission (asymptomatic)(S0) | 0 | 43
  Behavior - mild UC(S1): number analyzed (Participants) | 14 | 98
  Behavior - mild UC(S1) | 5 | 34
  Behavior - moderate UC(S2): number analyzed (Participants) | 14 | 98
  Behavior - moderate UC(S2) | 8 | 18
  Behavior - severe UC(S3): number analyzed (Participants) | 14 | 98
  Behavior - severe UC(S3) | 1 | 3
  Extraintestinal manifestations - Peripheral arthritis | 1 | 23
  Extraintestinal manifestations - Pyoderma gangrenosum | 0 | 2
  Extraintestinal manifestations - Aphthous ulcers | 0 | 1
  Extraintestinal manifestations - Primary sclerosing cholangitis | 0 | 1
  Extraintestinal manifestations - Osteoporosis | 0 | 2
  Extraintestinal manifestations - Anemia | 3 | 3
  Extraintestinal manifestations - Hematological alteration | 0 | 1
  Extraintestinal manifestations - Other | 10 | 70
Statistical Analysis 1: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Location of disease; Test type: Superiority; p = 0.2896, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 2: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Disease behavior; Test type: Superiority; p = 0.0006, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 3: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Extraintestinal manifestations: Peripheral arthritis; Test type: Superiority; p = 0.0890, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 4: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Extraintestinal manifestations: Pyoderma gangrenosum; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 5: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Extraintestinal manifestations: Aphthous ulcers; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 6: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Extraintestinal manifestations: Primary sclerosing cholangitis; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 7: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Extraintestinal manifestations: Osteoporosis; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 8: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Extraintestinal manifestations: Anemia; Test type: Superiority; p = 0.0752, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 9: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Extraintestinal manifestations: Hematological alteration; Test type: Superiority; p = 1.0000, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test
Statistical Analysis 10: Comparison: Moderate to Severe Ulcerative Colitis vs Mild to None Ulcerative Colitis; Extraintestinal manifestations: Other; Test type: Superiority; p = 0.1032, Chi-squared; p-value was obtained from Chi-square/Fisher's exact test

5. Secondary Outcome: Number of Participants With UC or CD Based on Inflammatory Bowel Disease (IBD) Therapies
Description: Number of participants will be reported based on the IBD therapies which include aminosalicylates, steroids, immunomodulators, immunosuppressants, biologics, antibiotics, probiotics, and surgeries. A participant can receive more than one IDB therapy.
Time Frame: From 3 years prior to Day 1 until Day 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 189
Participants
  Sulfasalazine (SSZ) | 1 | 1 | 6 | 14
  Mesalazine (5-ASA) | 20 | 25 | 36 | 140
  Olsalazine | 0 | 0 | 1 | 1
  Mesalazine extended release | 2 | 3 | 5 | 52
  Hydrocortisone | 4 | 3 | 5 | 17
  Prednisone | 18 | 23 | 19 | 77
  Prednisolone | 0 | 0 | 2 | 3
  Budesonide | 5 | 9 | 7 | 42
  Methylprednisolone | 0 | 0 | 1 | 0
  Azathioprine | 14 | 19 | 12 | 81
  6-mercaptopurine | 0 | 2 | 0 | 3
  Methotrexate | 4 | 3 | 1 | 0
  Infliximab | 13 | 9 | 9 | 46
  Adalimumab | 21 | 22 | 4 | 26
  Vedolizumab | 1 | 1 | 4 | 9
  Certolizumab | 4 | 1 | 0 | 0
  Golimumab | 0 | 0 | 2 | 3
  Ustekinumab | 13 | 8 | 2 | 1
  Metronidazole | 3 | 0 | 2 | 4
  Ciprofloxacin | 2 | 0 | 1 | 0
  Other | 14 | 3 | 11 | 44
  Salicylic derivatives + Immunosuppressants | 10 | 19 | 27 | 122
  Biologic therapy + Immunosuppressants | 12 | 14 | 1 | 4
  Salicylic derivatives + Immunosuppressants + Biologic therapy | 19 | 18 | 13 | 60

6. Secondary Outcome: Duration of IBD Therapies
Description: Time between the beginning of IBD therapy until the end of treatment or Day 1, whichever comes first. IBD therapies include aminosalicylates, steroids, immunomodulators, immunosuppressants, biologics, antibiotics, probiotics, and surgeries.
Time Frame: From 3 years prior to Day 1 until Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfill the study eligibility criteria. Number analyzed is the number of participants who had a complete duration from start to end date of therapy. Participants with incomplete or missing dates were not included in the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 189
months
  Sulfasalazine (SSZ): number analyzed (Participants) | 1 | 0 | 3 | 2
  Sulfasalazine (SSZ) | 0.2 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. |  | 33.3 [17.0 to 42.0] | 62.3 [40.3 to 84.3]
  Mesalazine (5-ASA): number analyzed (Participants) | 15 | 2 | 12 | 66
  Mesalazine (5-ASA) | 42.1 [3.7 to 111.1] | 34.3 [18.6 to 50.0] | 8.4 [0.2 to 347.2] | 54.3 [0.6 to 138.1]
  Mesalazine Extended release: number analyzed (Participants) | 1 | 0 | 0 | 0
  Mesalazine Extended release | 31.0 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. |  |  |
  Olsalazine: number analyzed (Participants) | 0 | 0 | 1 | 0
  Olsalazine |  |  | 60.0 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. |
  Hydrocortisone: number analyzed (Participants) | 2 | 1 | 6 | 10
  Hydrocortisone | 0.1 [0.10 to 0.13] | 0.1 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. | 0.2 [0.2 to 0.3] | 0.1 [0.0 to 0.3]
  Prednisone: number analyzed (Participants) | 10 | 7 | 18 | 58
  Prednisone | 5.0 [0.9 to 207.4] | 2.9 [1.1 to 83.9] | 1.6 [0.7 to 182.0] | 3.0 [0.1 to 148.5]
  Prednisolone: number analyzed (Participants) | 0 | 0 | 0 | 1
  Prednisolone |  |  |  | 3.2 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events.
  Budesonide: number analyzed (Participants) | 0 | 0 | 4 | 6
  Budesonide |  |  | 2.0 [1.3 to 12.4] | 2.8 [1.4 to 18.0]
  Azathioprine: number analyzed (Participants) | 8 | 4 | 15 | 39
  Azathioprine | 40.3 [2.7 to 111.1] | 38.6 [4.1 to 96.31] | 1.5 [0.06 to 153.5] | 45.5 [0.2 to 181.8]
  Methotrexate: number analyzed (Participants) | 2 | 0 | 1 | 0
  Methotrexate | 4.9 [3.8 to 6.0] |  | 0.7 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. |
  Metronidazole: number analyzed (Participants) | 1 | 0 | 3 | 2
  Metronidazole | 0.2 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. |  | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.3]
  Ciprofloxacin: number analyzed (Participants) | 0 | 0 | 1 | 0
  Ciprofloxacin |  |  | 0.2 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. |
  Infliximab: number analyzed (Participants) | 3 | 3 | 8 | 28
  Infliximab | 10.3 [0.8 to 17.0] | 62.3 [5.5 to 89.8] | 21.9 [3.1 to 73.4] | 14.2 [0.75 to 181.4]
  Adalimumab: number analyzed (Participants) | 6 | 3 | 1 | 20
  Adalimumab | 27.5 [0.19 to 125.2] | 34.27 [5.3 to 103.8] | 28.6 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. | 27.5 [0.1 to 125.2]
  Vedolizumab: number analyzed (Participants) | 0 | 0 | 0 | 1
  Vedolizumab |  |  |  | 9.0 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events.
  Ustekimumab: number analyzed (Participants) | 2 | 1 | 0 | 0
  Ustekimumab | 66.5 [50.4 to 82.6] | 1.0 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. |  |
  Certolizumab: number analyzed (Participants) | 3 | 0 | 0 | 0
  Certolizumab | 15.7 [3.9 to 132.0] |  |  |
  Golimumab: number analyzed (Participants) | 0 | 0 | 1 | 0
  Golimumab |  |  | 0.3 [NA to NA] — Minimum and Maximum range was not estimable due to insufficient number of participants with events. |
  Other:: number analyzed (Participants) | 2 | 0 | 12 | 16
  Other: | 23.8 [0.2 to 47.4] |  | 2.8 [0.1 to 128.2] | 4.5 [0.1 to 103.7]

7. Secondary Outcome: Percentage of Participants With UC or CD Based on Biologic-experience
Description: Percentage of participants who have experienced any biologic therapy (examples, infliximab, adalimumab, golimumab, ustekinumab, certolizumab) once or more than once according to medical history until the day 1. Percentages are rounded off to the nearest single decimal.
Time Frame: From 3 years prior to Day 1 until Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfill the study eligibility criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 189
percentage of participants | 72.0 | 61.5 | 33.0 | 33.8

8. Secondary Outcome: Percentage of Participants With UC or CD Who Have Not Responded Previously to Biologic Therapies
Description: Percentages are rounded off to the nearest single decimal.
Time Frame: From 3 years prior to Day 1 until Day 1
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 189
percentage of participants | 65.1 | 25.0 | 28.5 | 20.1

9. Secondary Outcome: Percentage of Participants With UC or CD Based on Reasons for Non-response to Previous Biologic Therapies
Description: Percentages are rounded off to the nearest single decimal.
Time Frame: From 3 years prior to Day 1 until Day 1
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 189
percentage of participants
  Poor effectiveness | 34.8 | 15.3 | 11.9 | 9.5
  Patient decision | 6.9 | 0 | 0 | 0
  Remission | 0 | 0 | 0 | 1.0
  Unknown | 0 | 0 | 4.7 | 2.1
  Patient poor adherence | 2.3 | 3.8 | 0 | 1.0
  Comorbidity | 0 | 0 | 0 | 0.5
  Adverse reaction | 4.6 | 0 | 0 | 3.7
  Patient access to treatment | 6.9 | 0 | 0 | 0.5
  Antibodies | 2.3 | 1.9 | 0 | 0.5
  Serum level of antidrug | 0 | 1.9 | 0 | 0
  Other | 6.9 | 1.9 | 11.9 | 1.0

10. Secondary Outcome: Number of Participants With UC or CD Introduced With IBD Treatment at Day 1
Description: The IBD treatment categories that have data for at least one participant are reported.
Time Frame: Day 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 189
Participants
  Sulfasalazine (SSZ) | 0 | 1 | 0 | 2
  Mesalazine (5-ASA) | 0 | 0 | 1 | 2
  Mesalazine extended release | 0 | 0 | 0 | 2
  Prednisone | 0 | 1 | 2 | 2
  Budesonide | 0 | 1 | 0 | 3
  Azathioprine | 0 | 1 | 1 | 0
  Infliximab | 0 | 0 | 0 | 1
  Adalimumab | 1 | 0 | 0 | 0
  Vedolizumab | 1 | 1 | 0 | 0
  Ustekinumab | 0 | 1 | 0 | 0
  Metronidazole | 0 | 0 | 1 | 0
  Ciprofloxacin | 0 | 0 | 1 | 0
  Other | 1 | 0 | 1 | 2

11. Secondary Outcome: Number of Participants With HBI >=8 or CDAI >=220 Points Versus HBI <8 or CDAI <220 Points Categorized Based on Socio-demographic, Clinical and Treatment-related Variables in CD Participants
Description: CDAI assessed clinical signs and symptoms: number of liquid stools, intensity of abdominal pain, general wellbeing, presence of comorbid conditions, use of antidiarrheal, physical examination and laboratory findings. Total score ranges from 0-600 points. Higher score indicates more severe disease. HBI score measures disease activity of CD based on 5 clinical parameters: general well-being, abdominal pain, number of liquid stools/day, abdominal mass, and complications. Total score is sum of individual parameters. Score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on number of liquid stools, where higher scores indicate more severe disease. Socio-demographic variables included age, sex, professional status, educational level, participant income. Clinical variables included duration and age at diagnosis, steroid dependence or refractoriness, family history, medical history and comorbidities, criteria used for diagnosis, calprotectin and EIM.
Time Frame: Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria. Data for participants with CD were reported.
Measure: Count of Participants; unit: Participants
Groups:
- Crohn's Disease: Participants diagnosed with CD were observed on Day 1 for cross-sectional evaluation of disease activity, treatment patterns, burden of disease and quality of life along with retrospective data collection for previous 3 years prior to Day 1 to assess the IBD treatments and use of other healthcare resources related with the management of CD.
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 95
Participants | 43

12. Secondary Outcome: Number of Participants With pMayo Score >=5 Versus pMayo Score <5 Categorized Based on Socio-demographic, Clinical and Treatment-related Variables in UC Participants
Description: Mayo score is composed of 4 categories (bleeding, stool frequency, physician assessment, and endoscopic appearance) rated from 0-3 that are summed into a total score ranging from 0-12. pMayo score consists of 3 sub scores: stool frequency, rectal bleeding, and physician global assessment of disease severity, each graded from 0 to 3. These scores were summed to give a total score range of 0 to 9; where higher scores indicating more severe disease. The pMayo score when compared with the full Mayo score and categorizes UC patients as being in remission (score of 0-2), having mild activity (pMayo of 3-4) or moderate to severe activity (pMayo >=5). Socio-demographic variables included age, sex, professional status, educational level, participant income. Clinical variables included duration and age at diagnosis, steroid dependence or refractoriness, family history, medical history and comorbidities, criteria used for diagnosis, calprotectin and extraintestinal manifestations (EIM).
Time Frame: Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria. Data for participants with UC were reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Ulcerative Colitis
Number analyzed (Participants) | 231
Participants | 42

13. Secondary Outcome: Mean Score of Components of 36-item Short Form Health Survey (SF-36) of UC or CD Participants
Description: SF-36 is a general quality of life (QoL)-questionnaire, which evaluates 8 health dimensions: physical functioning, bodily pain, role physical (limitations due to physical problems), role emotional (limitations due to personal or emotional problems), mental health, social functioning, vitality, and general health perceptions. Based on these 8 dimensions, two weighted scores were generated: the physical component summary (PCS) score and the mental component summary (MCS) score. Scores range between 0 and 100, with higher scores indicating a better quality of life. Mean score of each component (physical component and mental component) was reported.
Time Frame: Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants available for analysis for specified categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 188
score on a scale
  Physical Functioning | 64.2 (28.43) | 77.5 (24.10) | 71.1 (25.89) | 81.1 (22.97)
  Bodily Pain: number analyzed (Participants) | 43 | 52 | 42 | 187
  Bodily Pain | 52.7 (28.12) | 65.0 (27.90) | 57.5 (29.36) | 70.6 (26.09)
  Role Physical | 55.5 (28.87) | 62.9 (28.29) | 51.8 (26.63) | 69.9 (25.43)
  Role Emotional | 55.6 (28.51) | 62.2 (26.89) | 57.1 (28.07) | 70.6 (24.04)
  Mental Health: number analyzed (Participants) | 43 | 52 | 42 | 187
  Mental Health | 56.6 (20.43) | 60.9 (19.82) | 56.5 (22.62) | 64.8 (19.39)
  Social Functioning: number analyzed (Participants) | 43 | 52 | 42 | 187
  Social Functioning | 53.8 (29.19) | 66.6 (25.09) | 59.2 (28.70) | 69.7 (26.81)
  Vitality: number analyzed (Participants) | 43 | 52 | 42 | 187
  Vitality | 43.9 (20.30) | 53.7 (21.23) | 49.4 (22.55) | 57.2 (20.56)
  General Health | 43.4 (20.64) | 48.0 (23.59) | 43.4 (22.26) | 53.6 (23.62)

14. Secondary Outcome: Mean Total Score of Inflammatory Bowel Disease Questionnaire (IBDQ) of UC or CD Participants
Description: The IBDQ was a 32-item questionnaire that measured 4 dimensions: bowel function, emotional status, systemic symptoms, and social function. Within dimensions, each question presented seven possible answers/points. Each domain score was the sum of 8 responses each ranging from 1 to 7, where 1 indicated worst function and 7 the best. The sub-score ranged from 8 to 56 and thus the total score ranged from 32 to 224, where higher score indicating better quality of life.
Time Frame: Day 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 42 | 51 | 42 | 188
score on a scale | 144.8 (42.78) | 159.03 (36.00) | 140.2 (43.67) | 165.7 (33.85)

15. Secondary Outcome: Mean of Percentage of Total Work Impairment Assessed by Work Productivity and Activity Impairment Questionnaire (WPAI) in UC or CD Participants
Description: WPAI assessed the impact of IBD on work productivity and daily activities during the previous 7 days. The WPAI included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Employed participants were evaluated for this outcome measure. Mean total percentage of work impairment (absenteeism and presentisms) were reported in terms of hours.
Time Frame: The last 7 days prior to Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria. Overall number analyzed is the number of employed participants with data available for analysis for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of total work impairment
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 26 | 28 | 21 | 115
Percentage of total work impairment | 20.337 (19.2252) | 21.184 (21.4860) | 24.152 (15.6386) | 17.700 (19.6796)

16. Secondary Outcome: Mean of Percentage of Work Time Missed Assessed by WPAI in UC or CD Participants
Description: WPAI assessed the impact of IBD on work productivity and daily activities during the previous 7 days. The WPAI included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Employed participants were evaluated for this outcome measure. Mean work time missed (absenteeism) was reported.
Time Frame: The last 7 days prior to Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 26 | 28 | 21 | 118
percentage of work time missed | 19.873 (30.6995) | 17.285 (25.1336) | 9.798 (16.3332) | 10.590 (23.7578)

17. Secondary Outcome: Mean of Percentage of Impairment While Working Assessed by WPAI in UC or CD Participants
Description: WPAI assessed the impact of IBD on work productivity and daily activities during the previous 7 days. The WPAI included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Employed participants were evaluated for this outcome measure. Mean impairment while working (presentisms) was reported.
Time Frame: The last 7 days prior to Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage of Impairment
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 27 | 30 | 21 | 116
Percentage of Impairment | 33.3 (33.85) | 30.0 (30.40) | 29.5 (22.69) | 23.1 (25.92)

18. Secondary Outcome: Mean Percentage of Total Activity Impairment Assessed by WPAI in UC or CD Participants
Description: WPAI assessed the impact of IBD on work productivity and daily activities during the previous 7 days. The WPAI included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Unemployed participants only answered to questions related to employment status and regular activities impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Mean total activity impairment was reported.
Time Frame: The last 7 days prior to Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of total activity impairment
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 26 | 28 | 21 | 115
percentage of total activity impairment | 45.7 (35.87) | 33.1 (30.76) | 44.0 (30.45) | 27.4 (29.53)

19. Secondary Outcome: Percentage of Participants With UC or CD Who Quit Their Job Due to IBD and Unable to Return to Work
Description: Percentages are rounded off at the nearest single decimal.
Time Frame: Day 1
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 189
percentage of participants | 0 | 0 | 4.8 | 0

20. Secondary Outcome: Percentage of Participants With UC or CD Categorized Based on Healthcare Resources
Description: Healthcare resources included hospitalizations, medical appointments, imaging, and laboratory testing. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: From 3 years prior to Day 1 until Day 1
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 189
percentage of participants
  Hospital Admissions | 37.2 | 17.3 | 28.6 | 12.7
  Medical Appointments: IBD Specialist | 67.4 | 59.6 | 64.3 | 66.7
  Medical Appointments: Emergency Medical Appointment | 2.3 | 0 | 0 | 0
  Medical Appointments: Other Specialist | 4.7 | 0 | 2.4 | 4.2
  Imaging and Laboratory Testing | 60.5 | 61.5 | 52.4 | 67.2

21. Secondary Outcome: Total Direct Medical Cost for Participants With UC or CD
Description: A cost analysis of Ulcerative Colitis (UC) and Crohn's Disease (CD) was developed, classified by severity as mild and moderate-severe for each of the conditions. Direct medical costs were considered and included the following items: associated comorbidities, intestinal manifestations, surgical procedures, emergency visits, hospitalizations, medical appointments, follow-up studies, and previous pharmacological treatments; this was collected in the study including the number of participants and the proportion of them that presented the items studied. The total direct medical cost for all participants with each of the conditions was obtained, with the average 3-year cost per participant for UC and for CD multiplied by the number of all participants with UC and CD respectively. So, the values reported in the data table below represent the total direct cost for all participants with UC and CD respectively. The total direct cost was in Mexican Peso(MXN).
Time Frame: From 3 years prior to Day 1 until Day 1
Population: as for baseline characteristics
Measure: Number; unit: MXN
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 43 | 52 | 42 | 189
MXN | 16362506.13 | 12611636.50 | 9673667.75 | 33842289.53

22. Secondary Outcome: Indirect Cost for Participants With UC or CD
Description: A cost analysis of UC and CD was developed, classified by severity as mild and moderate-severe for each condition. Indirect cost was estimated by using number of hours missed from work (absenteeism) multiplied by average hourly labor cost including wages and benefits, to calculate average lost productivity cost per participant due to absenteeism during specified duration. Hours missed from work were assessed by Work Productivity and Activity Impairment Questionnaire: General Health (WPAI-GH) questionnaire, in which respondents answered 6 questions related to work productivity and impairment.The indirect medical cost for all participants with each of the conditions was obtained,with the average 3-year cost per participant for UC and for CD multiplied by the number of all employed participants with UC and CD respectively. So, values reported in data table below represent the indirect cost in totality for all employed participants with UC and CD respectively. The indirect cost is in MXN.
Time Frame: From 3 years prior to Day 1 until Day 1
Population: Enrolled Population Set included all participants who provided written informed consent and fulfilled the study eligibility criteria. Overall number of participants analyzed is the number of employed participants.
Measure: Number; unit: MXN
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
Number analyzed (Participants) | 27 | 30 | 21 | 120
MXN | 394402.91 | 276419.13 | 77869.29 | 458451.24

ADVERSE EVENTS:
Time Frame: Day 1
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Moderate to Severe Crohn's Disease | Mild to None Crohn's Disease | Moderate to Severe Ulcerative Colitis | Mild to None Ulcerative Colitis
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/52 | 0/42 | 0/189
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/52 | 0/42 | 0/189
Other Adverse Events (participants affected / at risk) | 0/43 | 0/52 | 0/42 | 0/189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT04873700/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT04873700/SAP_001.pdf